CLINICAL TRIAL: NCT04428034
Title: A Pilot Evaluation of Learning Skills Together: A Intervention to Teach Complex Care Skills to Caregivers of Persons Living With Alzheimer's Disease
Brief Title: Learning Skills Together Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC20200410H
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Family Caregiving; Complex Care; Self Efficacy; Intervention

STUDY DESIGN:
Intervention Model Description: A pre- and post-test design to test the Learning Skills Together program will be employed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learning Skills Together Intervention (Experimental): Participants in the Learning Skills Together program will begin their participation with a one-on-one phone call with an interventionist, who will ensure the participant is prepared to to attend the group sessions (e.g., familiar with videoconference technology) and will help the participant to set individual goals. The caregiver participant will then attend 4, group-based sessions lasting approximately 1.5 hours each, to learn about common complex care tasks managed by family caregivers to someone with mid-stage Alzheimer's disease, such as managing behavioral symptoms of dementia, incontinence, nutrition, transferring, medication management, and more. Sessions will integrate interactive activities, such as videos, case studies, and discussions. Approximately four weeks later, caregivers will be asked to attend a group reflection session to discuss application of what was learned and progress in meeting individual goals.
  Interventions: Behavioral: Learning Skills Together

INTERVENTIONS:
Behavioral: Learning Skills Together — Information provided in arm/group description.

SUMMARY:
The Learning Skills Together (LST) program is a synchronous web-based educational intervention developed to address the essential need for training to equip family caregivers to someone with mid-stage Alzheimer's disease to confidently provide complex care tasks.The purpose of this pilot study is to evaluate the feasibility of delivering LST, the program's acceptability to caregivers, and likelihood of effecting caregivers self-efficacy and mastery.

ELIGIBILITY:
Inclusion Criteria:

* Family member (including families of choice) to an individual living with Alzheimer's disease who has received a diagnosis from a physician
* Ages 18 and old
* Provides assistance with at least two instrumental activities of daily living or one activity of daily living
* Care recipient is described as being within mid-stage Alzheimer's Disease
* There are no plans to place the care recipient in a skilled nursing facility within the next 3 months

Exclusion Criteria:

* The caregiver is paid to provide care
* The caregiver does not have reliable access to a computer and internet
* The caregiver is unable to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible. Gender is self-reported. Participants may select "Male," "Female," and "Other" gender, and may select all responses that apply.
Enrollment: 41 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole L White, PhD, RN, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
De-identified study data will be made available to other researchers if requested.

REFERENCES:
- [Background] Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978 Mar;19(1):2-21. No abstract available. PMID 649936
- [Background] Pearlin LI, Mullan JT, Semple SJ, Skaff MM. Caregiving and the stress process: an overview of concepts and their measures. Gerontologist. 1990 Oct;30(5):583-94. doi: 10.1093/geront/30.5.583. PMID 2276631
- [Background] Chan EY, Glass G, Chua KC, Ali N, Lim WS. Relationship between Mastery and Caregiving Competence in Protecting against Burden, Anxiety and Depression among Caregivers of Frail Older Adults. J Nutr Health Aging. 2018;22(10):1238-1245. doi: 10.1007/s12603-018-1098-1. PMID 30498832
- [Background] Robertson, SM, Zarit, SH, Duncan, LG, Rovine, MJ, & Femia, EE. Family caregivers' patterns of positive and negative affect. Family Relations. 2007; 56(1): 12-23.

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to Intervention Completion
Arm/Group | Learning Skills Together Intervention
Started | 41
Attended at Least 2 Intervention Sessions in One Cohort | 35 (Forty-one (41) participants enrolled and completed the baseline survey. Of those who completed the baseline survey, three participants did not attend at least two sessions. Three participants started the intervention in one cohort but completed it in another (off-protocol).)
Completed | 35
Not Completed | 6
Not completed — Protocol Violation | 6
Period: 4-Week Follow Up Survey
Arm/Group | Learning Skills Together Intervention
Started | 35
Completed | 29
Not Completed | 6
Period: 8-Week Follow Up Survey
Arm/Group | Learning Skills Together Intervention
Started | 29
Completed | 27 (Of those 27 who completed the 8-week follow up survey, one participant skipped the 4-week follow up survey but completed the 8-week survey.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are described for the analysis population, which includes participants who were eligible according to initial criteria, but who also: 1) attended at least 2 program sessions and 2) completed the program in the same cohort (i.e., did not start in one cohort and complete "make up" sessions in the following cohort.
Arm/Group | Learning Skills Together Intervention
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: African American/Black | 3
  Race and Ethnicity: Asian | 3
  Race and Ethnicity: Caucasian/white | 19
  Race and Ethnicity: Hispanic | 10
Region of Enrollment [Number; unit: participants]
  United States | 35
Caregiver Competency [Mean (Standard Deviation); unit: units on a scale] — Measured using the Caregiver Competency Scale, a 3 item scale. Each scale has 5 responses: Never (0), to All of the time (5). Scores range from 3-15 with a lower score indicating less confidence in providing for relative's needs.
  units on a scale | 11.6 (2.6)
Caregiver Mastery [Mean (Standard Deviation); unit: units on a scale] — Measured using the Caregiver Mastery Scale, a 7 item scale which asks the participant the extent to which they feel they have control over various parts of their lives. Responses range from Strongly Disagree (1) to Strongly Agree (4). Range of scores are from 7-28, with a lower score showing that the caregiver believes they have less control.
  units on a scale | 16.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Competency
Description: This will be measured using the Caregiving Competence Scale. This measure includes 3-items pertaining to caregiver's confidence (e.g., "I feel confident that I am meeting the needs of my relative"). There are five response options to each statement ("Strongly Disagree" [1] to "Strongly Agree" [5]), such that scores may range from 3 to 15. A lower score indicates a lower level of confidence that the caregiver is meeting their relative's needs (i.e., higher scores are better). The outcome measure will use the average change score from baseline scores.
Time Frame: Change from baseline to 4 weeks post-intervention; and to 8 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learning Skills Together Intervention
Number analyzed (Participants) | 35
score on a scale
  4-Weeks Post-Intervention | 1.0 (1.6)
  8-Weeks Post-Intervention | 1.0 (2.2)

2. Primary Outcome: Change in Caregiver Mastery
Description: This will be measured using the Caregiver Mastery Scale. This 7-item scale asks participants the extent to which they feel they have control over various parts of their lives (e.g., "I have little control over the things that happen to me"). Participants may respond that they "Strongly Disagree (1) to Strongly agree (4) with each statement, such that scores range from 7 to 28. The lower the score, the less control the caregiver feels that they have control (i.e., higher scores are better). The mean score for this measure among caregivers to frail older adults was previously reported as 19.42 (SD 3.29), with Cronbach's alpha of 0.78. The outcome measure will use the average change score from baseline scores.
Time Frame: Change from baseline to 4 weeks post-intervention; and to 8 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learning Skills Together Intervention
Number analyzed (Participants) | 35
score on a scale
  4-Weeks Post-Intervention | 0.7 (2.3)
  8-Weeks Post-Intervention | 0.5 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year.
Arm/Group | Learning Skills Together Intervention
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Learning Skills Together Intervention (N=35)
Adverse Event: Identification of Severe Depression (Psychiatric disorders) | 3 (3) — This event pertains to caregivers who were identified during any measurement occasion as having severe depression. It is not known whether high depression scores were related to study participation.

LIMITATIONS AND CAVEATS:
Application of a. pre- and post-test design means that changes in self-efficacy cannot be attributed to the intervention alone

Results from this study are subject to selection bias given participant dropout between survey collection times

The small size of the analytic sample may have contributed to Type II error for some outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT04428034/Prot_SAP_000.pdf